CLINICAL TRIAL: NCT00880022
Title: Home-based Compression Therapy for Arm and Truncal Lymphedema in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Tactile Systems Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Sheila Ridner, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: supp930; NCT01097291 (obsolete NCT alias)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Arm Lymphedema; Truncal Lymphedema; Breast Cancer
Keywords: compression; Flexitouch; breast cancer; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm compression only (Active Comparator): Intervention of arm compression only by Flexitouch System
  Interventions: Device: Flexitouch System
- arm, trunk and chest compression (Experimental): Intervention of arm, trunk and chest compression by Flexitouch System
  Interventions: Device: Flexitouch System

INTERVENTIONS:
Device: Flexitouch System — ( 10 to 30 treatments depending on group assignment)

SUMMARY:
No studies have tested the potential benefit of the Flexitouch® truncal/chest garments on reducing truncal lymphedema in breast cancer survivors (BCS) or the theoretical added benefit of applying truncal/chest pneumatic compression therapy to open lymph channels in individuals who have only limb lymphedema or its impact on the trunk/chest. The purpose of this two-part study is to fill gaps related to: 1) the impact of the Flexitouch® System on truncal lymphedema, and 2) the therapeutic benefit of truncal /chest pneumatic compression therapy for arm lymphedema.

Hypotheses:

Part One: BCS with arm and truncal lymphedema. H1: Arm swelling (as measured by bioelectrical impedance & arm girth in cm) will be reduced after 10 sessions with the Flexitouch® System.

H2: Truncal swelling (as measured circumferentially) will be reduced after 10 sessions with the Flexitouch® System.

H3: The number, severity, and intensity, of physical and psychological symptoms (as measured by the Lymphedema Symptom Intensity and Distress Scale: Trunk and Arm) will be reduced after 10 sessions with the Flexitouch® System.

H4: Functional assessment scores (as measured by the Functional Assessment Screening Questionnaire [FASQ] will improve after 10 sessions with the Flexitouch® System.

Part Two: BCS with Arm Lymphedema H1: Arm volume (as measured by bioelectrical impedance & arm girth in cm) will be significantly reduced after one month of home use in participants using the Flexitouch® System (truncal, chest, and arm compression) when compared to those using the Flexitouch® System (arm compression only).

H2: Truncal measurements/volume (as measured circumferentially) will be less after one month of home use with the Flexitouch® System (truncal, chest, and arm compression) when compared to those using the Flexitouch® System (arm compression only).

H3: The number, severity, and intensity, of physical and psychological symptoms (as measured by Lymphedema Symptom Intensity and Distress Scale - Arm ) will be significantly reduced after one month of home use with the Flexitouch® System (truncal, chest, and arm garments) when compared to individuals using the Flexitouch® System (arm compression only) .

H4: Functional assessment scores (as measured by the FASQ) will be significantly higher after one month of home use with the Flexitouch® System (truncal, chest, and arm garments) when compared to individuals using the Flexitouch® System (arm compression only).

DETAILED DESCRIPTION:
Screening Procedures This study will have a three-phase screening process.

Phase One:

Participants will be screened either in person or via the telephone.

Phase Two:

If the person being interviewed is eligible and interested, study staff will obtain phone consent for a brief interview to obtain basic medical and treatment information and to share this information with the study doctor, who will write prescriptions for treatment based upon these data. After a prescription is obtained, study staff will contact participants by phone and schedule the on-site visit.

Phase Three:

Participants will come to the Vanderbilt University for measurement of arms and truncal assessment. Phase Three Screening informed consent will be obtained prior to any measurements. These measurements will serve as baseline entry into the study for those who meet criteria.

Baseline Interview All Participants: Once written informed consent is obtained, study staff will interview the participants to obtain demographic and treatment (lymphedema and breast cancer) history. Participants will complete symptom and quality of life forms.

Part One Study:

Dosage and Setting:

Participants will receive a total of 10 treatments, one hour per day for 10 days consecutively. Treatment One will be conducted under study staff supervision at VUSN or other Vanderbilt location. Treatments Two through Ten will be self-administered, at home, as this is an FDA approved at-home self-care device.

Study staff will make an at home visit for Treatment Two in order to observe the application and use of the device and to measure the participant's trunk and arms and examine arm and trunk.

Home Treatment One Observation and Measurement:

Physical Assessment/Measurement:

* Study staff will visually examine the affected and unaffected arms and truncal areas (collarbone to navel and small of back).
* Participants will be asked to sit at their dining table with arms extended to the side at shoulder height at shoulder level. A non-flexible tape will be used to measure girth at the metacarpal shaft of the hand and then, starting at the ulnar styloid, in 10 cm intervals to the shoulder. Each arm will be measured 2 times and the average used.
* Study staff will then measure the trunk twice at five locations.
* During bioimpedance: Study staff will assist the patient onto a bed or sofa and measure arm volume using bioelectrical impedance. Participants will be placed in a supine position with legs not touching one another. An alcohol pad will be used to prep each wrist next to the joint, the dorsal surface of each hand (1 cm proximal to the middle knuckle), and the dorsal surface of one foot (1 cm proximal to the joint of the second toe). These areas will be allowed to dry and lightly adhesive electrodes will be applied. Measurement of affected and unaffected arms will be conducted as directed by the computer software in each impedance device. This measurement will take less than five minutes. The leads and electrodes will then be removed.
* Study staff will weigh the participant twice and record the average.
* At the end of the treatment session, study staff will again measure the arms and trunk of the participant. Using the same procedures.

Treatment Observation:

Staff will observe for:

* Participants going to restroom, removing any compression garments, constrictive clothing/undergarments or foot coverings they are wearing, and to removing any jewelry prior to treatment.
* Participants changing into scrub suits.
* Use of treatment record checklist to set dials
* Participants resting in a supine position during treatment.
* Appropriate placement of garments.
* Pressures will be set at manufacturers recommended levels of compression using program UEO1/U1 and standard pressure (not intense pressure) only.
* Active time on the device approximately 60 minutes.
* Completion of treatment record checklist after treatment.
* Staff will correct any errors noted and educate as needed.

Measurement Visits (Between Treatment 5 and 6 (+ or - 1 treatment), and within 72 hrs after Treatment 10, Exit from Study):

Data Collection:

Physical Assessment/Measurement:

* Study staff will visually examine the affected and unaffected arms and truncal areas (collarbone to navel and small of back) and document findings on the Skin Checklist.
* Participants will be asked to sit at their dining table with arms extended to the side at shoulder height at shoulder level. A non-flexible tape will be used to measure girth at the metacarpal shaft of the hand and then, starting at the ulnar styloid, in 10 cm intervals to the shoulder. Each arm will be measured 2 times and the average used.
* Study staff will then measure the trunk at the five locations. During bioimpedance: Study staff will assist the patient to lay flat on a bed or sofa and staff will measure arm volume using bioelectrical impedance. Participants will be placed in a supine position with legs not touching one another. An alcohol pad will be used to prep each wrist next to the joint, the dorsal surface of each hand (1 cm proximal to the middle knuckle), and the dorsal surface of one foot (1 cm proximal to the joint of the second toe). These areas will be allowed to dry and lightly adhesive electrodes will be applied. Measurement of affected and unaffected arms will be conducted as directed by the computer software in each impedance device. This measurement will take less than five minutes. The leads and electrodes will then be removed .
* Study staff will weigh the participant twice and record the average.

Interview:

• Participants will complete the symptom and quality of life forms.

Part Two (Experimental and Control Groups)

Dosage and Setting:

Participants will receive a total of 30 treatments lasting up to approximately one hour per day for 30 days. Treatment One will be provided under study staff supervision . Treatments Two through Thirty will be self-administered, at home, as this is an FDA approved at-home self-care device.

Data Collection Initial On-Site Visit:

Physical Assessment/Measurement:

* Participants will be asked to void (for comfort during procedure), to remove any compression garments, constrictive clothing/undergarments, or foot coverings they are wearing, and to remove any jewelry.
* Participants will be asked to change into scrub suits.
* Participants will have their height (using a portable stadiometer) and weight (using a Pro-fit Electronic Scales) measured twice and the average will be recorded .

Treatment:

* Study staff will review the procedure in the manual for self-administration of the device and ask for participants to demonstrate their ability to apply the device and use the appropriate settings. Participants will view a video about the device.
* Participants will apply the Flexitouch® System garments (actual garment to be placed will be determined by randomization to experimental or control group) over and scrubs in the arm and trunk areas.
* Participants will rest supine on the massage table with their head on a pillow, if necessary, during treatment.
* For subjects randomized to the Experimental Group: Pressures will be set at manufacturers recommended levels of compression using the standard upper extremity program (UEO1/U1) and standard pressure (not intense pressure) only. Active time on the device will be approximately 60 minutes.
* For subjects randomized to the Control Group: pressures will be set at manufacturers recommended levels of compression using program for arm compression only (UE04/U4), chest will not receive compression, and standard (not intense pressure) only. Active treatment time for Group B patients will be approximately 40 minutes.
* Study staff will remain present during the treatment. Should a participant experience discomfort or request to stop the treatment, study staff will immediately turn off the device and remove the garments.
* At the end of the treatment session study staff will measure the arms and trunk.
* Trunk will be measured twice using a non-flexible tape.
* Bioelectrical Impedance: Study staff will assist the patient onto a non-metal massage table covered with clean linen and staff will measure arm volume using bioelectrical impedance. Participants will be placed in a supine position with legs not touching one another. An alcohol pad will be used to prep each wrist next to the joint, the dorsal surface of each hand (1 cm proximal to the middle knuckle), and the dorsal surface of one foot (1 cm proximal to the joint of the second toe). These areas will be allowed to dry and lightly adhesive electrodes will be applied. Measurement of affected and unaffected arms will be conducted as directed by the computer software in each impedance device. The leads and electrodes will then be removed and cleaned with an alcohol pad.
* Circumferential: With arms extended to the side and at shoulder level, a non-flexible tape will be used to measure girth at the metacarpal shaft of the hand and then, starting at the ulnar styloid, in 10 cm intervals to the shoulder.

Measurement Visits (After Treatment 14 (+or- 2 treatments) and within 72 hours after Treatment 30 (Exit from Study) :

Data Collection:

If the participant opts to come to Vanderbilt the measurement procedures for arms and weight will be the same as in the first onsite. If the visit takes place at-home the following procedures a will be used:

Physical Assessment/Measurement:

* Study staff will visually examine the affected and unaffected arms and truncal areas (collarbone to navel and small of back) and document findings on the Skin Checklist (Attachment C form 12).
* Participants will be asked to sit at their dining table with arms extended to the side at shoulder height. A non-flexible tape will be used to measure girth at the metacarpal shaft of the hand and then, starting at the ulnar styloid, in 10 cm intervals to the shoulder. Each arm will be measured 2 times and the average used.
* Study staff will then measure the trunk at the five locations noted on Attachment C form 11. Study staff will assist the patient onto a non-metal massage table covered with clean linen and staff will measure arm volume using bioelectrical.
* During bioimpedance: Study staff will ask the patient to lay flat on a bed or sofa and staff will measure arm volume using bioelectrical impedance. Participants will be placed in a supine position with legs not touching one another. An alcohol pad will be used to prep each wrist next to the joint, the dorsal surface of each hand (1 cm proximal to the middle knuckle), and the dorsal surface of one foot (1 cm proximal to the joint of the second toe). These areas will be allowed to dry and lightly adhesive electrodes will be applied. Measurement of affected and unaffected arms will be conducted as directed by the computer software in each impedance device. This measurement will take less than five minutes. The leads and electrodes will then be removed .
* Participants will be weighed twice and the average recorded.

Interview:

• Participants will complete the symptom and quality of life forms.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals at least six months post- surgery and/or radiation treatment for breast cancer
2. At least 21 years of age
3. Lymphedema in one arm subsequent to breast cancer treatment with coexisting truncal swelling ** (Part One) and *lymphedema in one arm subsequent to breast cancer treatment without coexisting truncal swelling (Part Two)
4. Willing and able to drive to the study site as needed
5. Currently not using a compression pump or undergoing manual lymphatic drainage by a therapist

Exclusion Criteria:

1. Actively undergoing or less than six months post intravenous chemotherapy or radiation therapy
2. Individuals with congestive heart failure, chronic/acute renal disease, cor pulmonal, nephrotic syndrome, nephrosis, liver failure or cirrhosis, pulmonary edema, thrombophlebitis, deep vein thrombosis, infection of any kind and inflammation (redness) in the trunk or arms
3. History of bilateral breast cancer
4. Metastatic cancer
5. Inability to stand upright
6. Metal implants that would interfere with bioimpedance measurement equipment
7. Pregnancy
8. Pacemaker and internally implanted defibrillators

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila H Ridner, Phd, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt Univeristy, Nashville, Tennessee, United States

REFERENCES:
- [Result] Ridner SH, Murphy B, Deng J, Kidd N, Galford E, Dietrich MS. Advanced pneumatic therapy in self-care of chronic lymphedema of the trunk. Lymphat Res Biol. 2010 Dec;8(4):209-15. doi: 10.1089/lrb.2010.0010. PMID 21190493
- [Result] Ridner SH, Murphy B, Deng J, Kidd N, Galford E, Bonner C, Bond SM, Dietrich MS. A randomized clinical trial comparing advanced pneumatic truncal, chest, and arm treatment to arm treatment only in self-care of arm lymphedema. Breast Cancer Res Treat. 2012 Jan;131(1):147-58. doi: 10.1007/s10549-011-1795-5. Epub 2011 Sep 30. PMID 21960113

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm Compression Only; Arm, Trunk and Chest Compression: Participants received a total of 30 treatments lasting up to approximately one hour per day for 30 days. Treatment One was provided under study staff supervision. Treatments Two through Thirty were self-administered, at home.
Period: Overall Study
Arm/Group | Arm Compression Only | Arm, Trunk and Chest Compression
Started | 23 | 24
Completed | 21 | 21
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm Compression Only | Arm, Trunck and Chest Compression | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (9.3) | 52.2 (8.6) | 55.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Arm Volume at End of Study
Description: measured by tape and then volume was calculated.
Time Frame: end of scheduled treatments-day 30 of treatment
Population: Study withdrawals were not included.
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Arm Compression Only | Arm, Trunck and Chest Compression
Number analyzed (Participants) | 21 | 21
ml | 2376.52 [1934.68 to 2622.99] | 2539.93 [2168.28 to 3295.97]

2. Secondary Outcome: Symptom Improvement
Description: Lymphedema Symptom and Intensity Scale-Arm measures 30 symptoms yes no over the past 7 days . Total yes items added for number of symptoms.
Time Frame: Before first treatment and end of all treatments
Population: Number of participant symptoms
Measure: Median (Inter-Quartile Range); unit: Number of participant symptoms
Groups:
- Arm Compression Only: Compression in Arm only
- Arm, Trunk and Chest Compression: Compression in arm, trunk and chest compression
Arm/Group | Arm Compression Only | Arm, Trunk and Chest Compression
Number analyzed (Participants) | 21 | 21
Number of participant symptoms
  Baseline | 12.0 [7.5 to 16.0] | 15.0 [9.5 to 20.0]
  End of Treatment | 6.0 [4.0 to 11.5] | 10.0 [6.0 to 17.5]

ADVERSE EVENTS:
Arm/Group | Arm Compression Only | Arm, Trunck and Chest Compression
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No